CLINICAL TRIAL: NCT05852899
Title: Evaluation of Preoperative Risk Factors in Prediction of ICU Admission in Children, An Observational Prospective Study
Brief Title: Evaluation of Preoperative Risk Factors in Children
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, tugba yesilyurt dogu, medical doctor, Istanbul University - Cerrahpasa
Other Study IDs: 144674
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia Morbidity; Preterm Birth; Difficult or Failed Intubation
Keywords: ASA-PS; surgical risk; risk assessment; preoperative; prediction of icu admission
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. The investigators aimed to make a more advanced risk assessment in predicting preoperative intensive care unit admission in pediatric patients.
2. The investigators aimed to better define the pediatric patient population and identify preoperative risk factors in detail in order to reduce perioperative complications.

DETAILED DESCRIPTION:
The aim of this study was to evaluate preoperative risk factors and determine their efficacy in predicting ICU admission after emergency or elective surgery in pediatric patients of all age groups. To achieve this aim, data such as gender, age, height, weight, history of prematurity, post-conceptional week, ASA PS score, accompanying systemic diseases, history of previous anesthesia, history of emergency or elective surgery, tumor surgery, chemotherapy and radiotherapy, surgical risk classification, difficult airway will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Children under the age of 18 who will have an operation in the pediatric surgery operating room.

Exclusion Criteria:

* Children who are scheduled for surgery in pediatric surgery room but are hospitalized in the intensive care unit.(Children admitted directly from the intensive care units to the operating rooms)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under the age of 18 who will have an operation in the pediatric surgery operating room at Cerrahpasa Medical Faculty
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
ASA-PS | Preoperative visit period ( 20 minutes)
  The American Society of Anesthesiologists (ASA) physical status preoperative risk assesttment
Postoperative PICU admission | postoperative follow-up ( in 72 hours)
  Number of participants of Postoperative Pediatric Intensive Care Unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Yesilyurt Dogu, MD, Principal Investigator — Istanbul University- Cerrahpaşa (IUC); Pinar Kendigelen, MD, Study Director — Istanbul University- Cerrahpaşa (IUC); Ayse Cigdem Tutuncu, MD, Study Chair — Istanbul University- Cerrahpaşa (IUC)
Locations (1):
- Tuğba Yeşilyurt Doğu, Istanbul, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
ASA PS, surgical risk, demographic datas, preoperative hemoglobin, preoperative SpO2.